CLINICAL TRIAL: NCT02807883
Title: Blinatumomab Maintenance Following Allogeneic Hematopoietic Cell Transplantation for Patients With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0576; NCI-2016-01182 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; ALL; B-lineage Acute Lymphoblastic Leukemia; Malignant neoplasms stated as primary lymphoid haematopoietic; Blinatumomab; Blincyto; Post allogeneic stem cell transplant
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Blinatumomab (Experimental): Blinatumomab as continuous intravenous infusion at dose of 28 µg/24 hours over 4 weeks followed by 2 week treatment-free period for 6-week treatment cycle; 4 cycles of blinatumomab at 3, 6, 9, and 12 months following hematopoietic cell transplantation (HCT).
  Interventions: Drug: Blinatumomab; Procedure: Hematopoietic Cell Transplantation

INTERVENTIONS:
Drug: Blinatumomab — Participants receive Blinatumomab as continuous intravenous infusion at a dose of 28 µg/24 hours over 4 weeks followed by a treatment-free period of 2 weeks, defined as one 6-week treatment cycle. In the first induction cycle, the initial dose of Blinatumomab is 9 µg/day for the first 7 days of treatment which then will be escalated (dose step) to 28 µg/day starting on day 8 (week 2) through day 29 (week 4). For all subsequent cycles, 28 µg/day is the dose for all 4 weeks of continuous treatment. Participants receive 4 cycles of blinatumomab at 3, 6, 9, and 12 months following hematopoietic cell transplantation (HCT).
  Other Names: Blincyto
Procedure: Hematopoietic Cell Transplantation — Hematopoietic progenitor cell infusion
  Other Names: HCT

SUMMARY:
You are being asked to take part in this study because you either had Ph positive B-lineage acute lymphoblastic leukemia (ALL) or still have a small amount of the disease and recently received an allogeneic stem cell transplant (cells from someone else).

The goal of this clinical research study is to learn if blinatumomab in patients who have had an allogeneic stem cell transplant can help to control ALL or prevent ALL from coming back in patients who either have a small amount of ALL or have had ALL in the past. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Study Drug Administration:

Every study cycle will be 6 weeks. You may receive up to 4 cycles of blinatumomab. Each cycle will start around 3, 6, 9, and 12 months after your stem cell transplant.

In each cycle, you will receive blinatumomab as a continuous infusion by vein for 4 weeks, followed by a 2 week "rest period" during which you will not receive blinatumomab.

You will need to remain in the hospital for the first 2 cycles so that you can be checked on for side effects.

Length of Study:

You may receive blinatumomab for up to 1 year. You will no longer be able to receive the study drug if the disease comes back (if you do not have ALL), if the disease gets worse (if you have a small amount of ALL), if intolerable side effects occur, or if you are unable to follow study directions.

Study Visits:

Before each cycle:

* You will have a physical exam. As part of the physical exam, you will be checked for graft versus host disease (GVHD, when transplanted donor tissue attacks the tissues of the recipient's body).
* Blood (about 4 tablespoons) will be drawn to learn the effectiveness of the stem cell transplant.
* You will have a bone marrow biopsy and aspiration to check the status of the disease and for cytogenetic testing.

Once a week during each cycle, blood (about 4 tablespoons) will be drawn for routine tests.

End of Study Visit:

About 2 weeks after your last dose of blinatumomab:

* You will have a physical exam.
* Blood (about 4 tablespoons) will be drawn to learn the effectiveness of the stem cell transplant.
* You will have a bone marrow biopsy and aspiration to check the status of the disease and for cytogenetic testing.

This is an investigational study. Blinatumomab is FDA approved and commercially available for the treatment of Philadelphia chromosome (Ph) negative B-ALL that has returned after treatment. Its use in patients with Ph positive B-lineage ALL is investigational.

Up to 30 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 1-70 years of age.
2. Patients with B-lineage ALL in a) hematologic complete remission (CR) beyond CR1 at time of transplant; patients beyond CR1 or with primary induction failure may be without minimal residual disease, b) any residual disease defined by positive flow >0.01%, detection of BCR-ABL transcript by PCR with a sensitivity of 1/10,000, or detection of the t(9;22) translocation in any metaphases by cytogenetics at time of transplant, or presence of the MLL gene.
3. Received an allogeneic HCT within the last 100 days. Enrollment within 30-100 days after transplant, and after adequate recovery of counts defined as ANC >/= 0.5 x 10^9/L without daily use of myeloid growth factor and platelet > 20 x 10^9/L without platelet transfusion within 1 week, and adequate organ function to receive blinatumomab defined as creatinine clearance greater than 30 ml/min, ALT/AST < 5 x ULN and serum bilirubin < 3 x ULN.
4. Performance status of 0, 1, or 2. Karnofsky (or Lansky for subjects < 16 years old) performance status >/= 50.

Exclusion Criteria:

1. Relapsed ALL defined as >5% malignant blasts in bone marrow or peripheral blood.
2. Active GVHD requiring systemic steroid therapy. Medications for GVHD prophylaxis are acceptable.
3. Systemic steroid therapy unless for physiologic replacement
4. Uncontrolled disease/infection as judged by the treating physician
5. Active ALL in the central nervous system (CNS), as defined by >/= 5 leukocytes per microL with identifiable blast cells in the CSF, and/or the presence of cranial-nerve palsies
6. Pregnant or nursing women

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Partow Kebriaei, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Gaballa MR, Banerjee P, Milton DR, Jiang X, Ganesh C, Khazal S, Nandivada V, Islam S, Kaplan M, Daher M, Basar R, Alousi A, Mehta R, Alatrash G, Khouri I, Oran B, Marin D, Popat U, Olson A, Tewari P, Jain N, Jabbour E, Ravandi F, Kantarjian H, Chen K, Champlin R, Shpall E, Rezvani K, Kebriaei P. Blinatumomab maintenance after allogeneic hematopoietic cell transplantation for B-lineage acute lymphoblastic leukemia. Blood. 2022 Mar 24;139(12):1908-1919. doi: 10.1182/blood.2021013290. PMID 34914826
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruitment from August 2016 to June 2020 at MD Anderson Cancer Center
Pre-assignment Details: 23 participants signed consents, 2 participants withdrew before treatment.
Period: Overall Study
Arm/Group | Blinatumomab
Started | 23
Completed | 21
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Blinatumomab
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
  Mexico | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Toxicities
Description: Participants with treatment-related toxicities attributable to Blinatumomab. Toxicities defined as any 1) grade 3-4 acute GVHD greater than 30%, 2) secondary graft failure >30%, or 3) nonrelapse mortality (NRM) within one cycle of Blinatumomab.
Time Frame: 30 days from the first cycle
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 21
Participants | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Number of participants with progression free survival from the date of allogeneic HCT to the date of disease progression or death. (Progression is defined as more than 5% blast in the peripheral blood or bone marrow biopsy.)
Time Frame: From last treatment cycle, assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 21
Participants | 15

3. Secondary Outcome: Overall Survival (OS)
Description: Number of participants in the study who are alive and disease free up to 1 year.
Time Frame: From last treatment cycle, assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 21
Participants | 18

ADVERSE EVENTS:
Time Frame: Adverse event were collected up to 30 days from the last treatment cycle.
Arm/Group | Blinatumomab
All-Cause Mortality (participants affected / at risk) | 3/23
Serious Adverse Events (participants affected / at risk) | 5/23
Other Adverse Events (participants affected / at risk) | 20/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=23)
Low granulocyte (Blood and lymphatic system disorders) | 4
Secondary graft failure (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=23)
Abdominal pain (Gastrointestinal disorders) | 1
ALK increased (Investigations) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1
ALT increased (Investigations) | 9
Anemia (Investigations) | 1
Anxiety (Psychiatric disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
AST increased (Investigations) | 5
Bacterial (Infections and infestations) | 1
CD OTH (Cardiac disorders) | 1
Chest pain (Cardiac disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 2
Diarrhea (Gastrointestinal disorders) | 7
Dysrhythmia (Cardiac disorders) | 1
Dizziness (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Dry eye (Eye disorders) | 1
Fatigue (General disorders) | 4
Fever (General disorders) | 3
Headache (Nervous system disorders) | 3
Flu like syndrome (General disorders) | 1
Insomnia (Psychiatric disorders) | 3
Low granulocyte (Blood and lymphatic system disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 7
Low platelet (Investigations) | 4
NE COR (General disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Oral mucositis (Gastrointestinal disorders) | 1
Thromboembolic event (Vascular disorders) | 2
Viral (Infections and infestations) | 2
Secondary graft failure (Blood and lymphatic system disorders) | 1
Tremor (Nervous system disorders) | 1
Wbc decreased (Investigations) | 12
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT02807883/Prot_SAP_000.pdf